CLINICAL TRIAL: NCT05453630
Title: Colonoscopy Outreach for Rural Communities Aim 2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Alison Cole, Associate Professor, School of Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: STUDY00014807; 1R01CA254515-01 (NIH)
Record Dates: First submitted 2022-07-06; First posted 2022-07-12 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-07

CONDITIONS: Colorectal Cancer
Keywords: colorectal cancer; patient navigation; colonoscopy; FIT; fecal immunochemical test; immunochemical fecal occult blood test; implementation effectiveness; colorectal cancer screening
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Patient Navigation

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient Navigation Intervention (Experimental): Patients randomized to this arm will receive language-concordant patient navigation from a trained navigator, over the phone and via text and email, to assist patients to complete colonoscopy to screen for colorectal cancer.
  Interventions: Behavioral: Patient Navigation
- Standard of Care Control (Other): Participants randomized to this arm will receive an educational brochure about the importance of colonoscopy to screen for colorectal cancer.
  Interventions: Behavioral: Usual Care Control

INTERVENTIONS:
Behavioral: Patient Navigation — Patients will receive navigation from a trained lay navigator at a community-based nonprofit organization that supports access to high quality healthcare. The patient navigator will work with patients to schedule their colonoscopy and identify, explore, and overcome barriers. They will educate patients about the colonoscopy procedure and preparation, provide resources, and coach and motivate patients.
  Arms: Patient Navigation Intervention
Behavioral: Usual Care Control — Educational brochure about colonoscopy
  Arms: Standard of Care Control

SUMMARY:
This study aims to test the effectiveness of a remotely-delivered patient navigation program for increasing colonoscopy completion for colorectal cancer screening, among rural populations. The study will partner with geographically disparate primary care organizations to recruit patients aged 45-75 to the study. The patient navigation program will be delivered through a community organization. This project is critical in advancing our knowledge of the effectiveness of patient navigation for increasing colonoscopy in this patient population as well as for understanding factors that can support long term implementation and sustainability of effective interventions.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) is a leading cause of cancer death in the United States and its burden is greater in rural and low-income communities. Failure to complete recommended colonoscopy contributes to later-stage CRC diagnosis and worse CRC outcomes, which means timely and successful colonoscopy is a key opportunity to reduce CRC mortality. Using a Type 1 Hybrid Implementation-Effectiveness design, we will randomize 480-600 subjects from 6-8 primary care clinical organizations in a randomized controlled trial (RCT) to accomplish the following:

* Test the effectiveness of a patient navigation program, remotely-delivered by a community-based organization, for increasing colonoscopy completion rates for colorectal cancer screening among rural patients.
* Assess implementation and sustainability of the patient navigation program from the perspectives of both community and clinical stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* Aged 45-76.25 on the date of their referral for colonoscopy
* Referred for colonoscopy as part of colorectal cancer screening in the last 3 months. This includes patients referred for colonoscopy after an abnormal stool screening test (e.g., FIT/FOBT/Cologuard) and patients referred for colonoscopy as a primary screening test for colorectal cancer.

Exclusion Criteria:

* Deceased
* Colonoscopy procedure since colonoscopy referral
* Colonoscopy procedure scheduled less than or equal to 7 days from study enrollment date
* Colonoscopy procedure scheduled more than 9 months from colonoscopy referral date (if known at enrollment)
* Have diagnosis or past history of total colectomy or colorectal cancer (malignant neoplasm) at any time
* Has hospice
* Aged 66 and older living long-term in an institution for more than 90 consecutive days during the year prior to the query

Ages: 45 Years to 915 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 527 (Actual)
Dates: Start 2022-06-16 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-07-15 (Actual)

PRIMARY OUTCOMES:
Number of participants who complete colonoscopy within 1 year of the colonoscopy referral | 1 year

SECONDARY OUTCOMES:
Number of participants who complete colonoscopy within 6 months of the colonoscopy referral | 6 months
Time to completion of colonoscopy or end of follow-up after the colonoscopy referral | 1 year
Number of participants who complete colonoscopy within 9 months of the colonoscopy referral | 9 months
Number of participants who have completed colonoscopies with adequate preparation | 1 year
Number of participants who have colonoscopies with cecal intubation | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Allison M Cole, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- University of Washington, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Keppel GA, Ike B, Leroux BG, Ko LK, Osterhage KP, Jacobs JD, Cole AM. Colonoscopy Outreach for Rural Communities (CORC): A study protocol of a pragmatic randomized controlled trial of a patient navigation program to improve colonoscopy completion for colorectal cancer screening. Contemp Clin Trials. 2024 Jun;141:107539. doi: 10.1016/j.cct.2024.107539. Epub 2024 Apr 12. PMID 38615750